CLINICAL TRIAL: NCT04493021
Title: Evaluation of the Dermal Cooling System for the Enhanced Treatment of Benign Pigmented Lesions and Common Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R2 Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-20-001
Record Dates: First submitted 2020-07-26; First posted 2020-07-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with Dermal Cooling System (Experimental): Dermal Cooling System will be used in all eligible subjects.
  Interventions: Device: Dermal Cooling System

INTERVENTIONS:
Device: Dermal Cooling System — Controlled localized cooling will be applied to benign pigmented lesions using the Dermal Cooling System

SUMMARY:
The purpose of this study is to evaluate the Dermal Cooling System for lightening of benign pigmented lesions and to assess additional cosmetic benefits.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label study to evaluate the effectiveness of the Dermal Cooling system to reduce pigmentation in benign pigmented lesions and to determine if additional cosmetic benefits are achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has one or more benign pigmented lesions (e.g., solar lentigines, freckles, seborrheic keratosis), in an area suitable for treatment.
3. Subject is willing to have up to 40 treatment sites treated per treatment session depending on the size and nature of the lesions identified.
4. Subject is willing to have digital photographs taken of the treatment area and agrees to use of photographs for presentation, educational, or marketing purposes.
5. Subject is willing to cover treated area or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area for the duration of the study, including the follow-up period, if requested.
6. Subject has read and signed a written informed consent form.
7. Subject is willing to comply with adjuvant topical regimen, as applicable. -

Exclusion Criteria:

1. Physician prescribed medical or surgical treatment, or use of over-the-counter products to alter skin color, in the area of intended treatment in the previous 6 months (e.g., hydroquinone, corticosteroids, laser surgery)
2. Use of products containing glycolic acids, retinol, salicylic acid within the previous 2 weeks
3. Use of Accutane within the previous 6 months
4. Artificial tanning in the area of intended treatment within 1 month (e.g., spray, lotion, tanning bed) or intention to use artificial tanning within the follow-up period
5. Scars or tattoos in the location of the treatment sites
6. History of melasma, vitiligo, eczema, or psoriasis in the area of treatment
7. History of melanoma
8. Subject is pregnant or intending to become pregnant during the study period
9. Subject is lactating or has been lactating in the past 6 months
10. Known history of illness or adverse reaction to cold insult (e.g., cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria, Reynaud's disease.
11. History of abnormal wound healing or abnormal scarring
12. Inability or unwillingness to comply with the study requirements.
13. Current enrollment in a clinical study of any other unapproved investigational drug or device.
14. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Improvement in the appearance of the treated areas as assessed by Investigator assessment. | 2-Month Follow-up visit
  Investigator assessment using Global Aesthetic Improvement Scale (GAIS); graded from "4" (very much improved") to "0" (worse).
Safety of the treatment | Up to 12 months
  Determined by incidence of device-or procedure-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Andre Bonnett, MD, Principal Investigator — Sculptology
Locations (1):
- Sculptology, Pleasanton, California, United States